CLINICAL TRIAL: NCT07106723
Title: A Clinical Study of the Safety and Efficacy of Autologous Hematopoietic Stem Cell Transplantation in Combination With CD7-CART in the Treatment of CD7+ T-Cell Lymphoma
Brief Title: Clinical Study of the Safety and Efficacy of ASCT Combined With CD7-CART in the Treatment of CD7+ TCL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Hebei Taihe Chunyu Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025051
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: CD7 Positive; T - Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell

STUDY DESIGN:
Intervention Model Description: ASCT conbined with CD7-CART
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ASCT conbined with CD7-CART. (Experimental)
  Interventions: Drug: ASCT+CD7-CART

INTERVENTIONS:
Drug: ASCT+CD7-CART — Intravenous infusion of CD7-CART 3 days after ASCT

SUMMARY:
To evaluate the safety and efficacy of autologous hematopoietic stem cell transfer (ASCT) combined with CD7-CART in the treatment of CD7+ TCL

ELIGIBILITY:
Inclusion Criteria:

1. With the subject's consent and having signed the informed consent form, willing and capable of adhering to the planned visits, study treatment, laboratory tests and other trial procedures;
2. Age 18 to 65 years old, both male and female;
3. Confirmed as T-cell non-Hodgkin's lymphoma type (including T-lymphoblastic lymphoma/leukemia) according to the World Health Organization's classification of hematopoietic and lymphoid tissue tumors (2022), and meeting one of the following three conditions: 1) Newly diagnosed with high-risk factors, such as Ann Arbor stage III/IV, large mass, bone marrow invasion, central nervous system (CNS) invasion, ETP phenotype, RAS activating mutation, TP53 deletion/mutation, etc., as assessed by the investigator; 2) Not achieving PR or better response after induction and consolidation therapy; 3) Patients not considered for allogeneic hematopoietic stem cell transplantation;
4. Confirmed as tumor cells expressing CD7 by histopathology and/or cytology at the time of screening;
5. With appropriate organ function: 1) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 times the upper limit of normal (ULN), if the investigator determines that the abnormal ALT and AST are due to the disease (such as liver infiltration or bile duct obstruction), the indicators can be relaxed to ≤ 5 times ULN; 2) Total serum bilirubin ≤ 2 times ULN, except for patients with Gilbert's syndrome; patients with Gilbert's syndrome and total bilirubin ≤ 3 times ULN and direct bilirubin ≤ 1.5 times ULN can be included; 3) Serum creatinine clearance rate ≥ 30 mL/min; 4) International normalized ratio (INR) ≤ 1.5 times ULN, and activated partial thromboplastin time (aPTT) ≤ 1.5 times ULN; 5) Possessing the minimum level of lung reserve, defined as ≤ grade 1 dyspnea (CTCAE v5.0) and non-oxygen-dependent blood oxygen saturation ≥ 92%; 6) Left ventricular ejection fraction ≥ 50% by echocardiography; no clinically significant abnormal electrocardiogram findings; no clinically significant pericardial effusion and pleural effusion.
6. Women of childbearing age have a negative blood/urine pregnancy test within 7 days before infusion. Any male and female patients with fertility must agree to use effective contraceptive methods throughout the study and for at least 2 years after the administration of study treatment.

   -

Exclusion Criteria:

Subjects with one or more of the following are not eligible for this study:

1. History of allergy to any of the components in the cell product;
2. Severe cardiac disease, including but not limited to: Myocardial infarction, cardiac angioplasty, or stenting within 6 months prior to signing the ICF; unstable angina; severe cardiac arrhythmias; History of severe non-ischemic cardiomyopathy; Congestive heart failure (New York Heart Association [NYHA] Class III or IV), NYHA score listed in Appendix II
3. Have a history of autologous/allogeneic hematopoietic stem cell transplantation;
4. stroke or seizure within 6 months prior to signing the ICF;
5. Have autoimmune diseases, immunodeficiencies or other diseases that require immunosuppressant treatment;
6. Within 3 years prior to signing the ICF, have malignancies other than T-cell hematologic tumors, except for adequately treated carcinoma in situ of the cervix, basal cell or squamous epithelial cell skin cancer, localized prostate cancer after radical resection, carcinoma in situ of the duct in situ after radical resection, carcinoma in situ of other sites one year after radical resection, and there has been no treatment during the screening period and there is no sign of recurrence;
7. presence of uncontrolled active infection;
8. Unstable systemic diseases judged by the investigator: including but not limited to severe hepatic, renal or metabolic diseases requiring drug treatment;
9. Any of the following within 4 weeks prior to lymphocyte collection:

The DNA detection value of hepatitis B virus (HBV) in peripheral blood was higher than the lower limit of detection; Positive for hepatitis C virus (HCV) antibody and positive for peripheral HCV-RNA; positive for human immunodeficiency virus (HIV) antibodies; positive for syphilis antigen or antibody; Positive for CMV-DNA (10) application of prednisone (or equivalent amounts of other corticosteroids) in excess of 5mg/day within 1 week prior to lymphocyte collection; (11) Have used any CAR-T cell products or other genetically modified T-cell therapies; (12) Received CD7-targeted therapy; (13) History of live vaccination within 4 weeks prior to signing the ICF; (14) Have a history of alcoholism, drug abuse, or mental illness; (15) Other situations that the investigator considers unsuitable to participate in this study.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2029-01-07 (Estimated); Study Completion 2030-01-07 (Estimated)

PRIMARY OUTCOMES:
PFS rate at 1 year after ASCT conbined with CD7-CART | at 1 year after ASCT conbined with CD7-CART
Incidence and Severity of Adverse Events after ASCT conbined with CD7-CART | during 2 years after ASCT conbined with CD7-CART
  Refer to irAE grading standard

SECONDARY OUTCOMES:
Duration of Response (DOR) | during 2 years after ASCT conbined with CD7-CART
  Time from first response evaluated by investigator to disease progression or death from any cause
Progression-free Survival (PFS) | during 2 years after ASCT conbined with CD7-CART
MRD negetive rate | at 3 or 6 month after ASCT conbined with CD7-CART
Time to Response (TTR) | during 2 years after ASCT conbined with CD7-CART
  Time from CD7-CART infusion to first documentation of response evaluated by investigators
Overall Survival (OS) | during 2 years after ASCT conbined with CD7-CART
Cmax | during 3 month after ASCT conbined with CD7-CART
  the peak CARgene copy number in peripheral blood
Tmax | during 3 month after ASCT conbined with CD7-CART
  time to reach the peak of CARgene copy number in peripheral blood
AUC(0-28d) | during 28 days after ASCT conbined with CD7-CART
  area under curve of CARgene copy number in peripheral blood
Tlast | during 1 year after ASCT conbined with CD7-CART
  duration of existence of CARgene copy number in peripheral blood

CONTACTS AND LOCATIONS:
Locations (1):
- Blood Disease Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China